CLINICAL TRIAL: NCT04054505
Title: Quantitative Analysis of Clinical Data for the Effectiveness of a Nutraceutical in Raising Circulating Serum Vitamin, Mineral and Amino Acid Levels in Patients.
Brief Title: Effectiveness of a Nutraceutical in Raising Circulating Serum Vitamin, Mineral and Amino Acid Levels in Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optimal Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: EZ102018
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Vitamin Deficiency
MeSH Terms: conditions — Avitaminosis

STUDY DESIGN:
Intervention Model Description: Triple blind
Who Masked: Participant, Care Provider, Investigator
Masking Description: Unmarked plan packet
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- Vitamin A (Active Comparator): Rise or fall of Vitamin A after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- Vitamin E (Active Comparator): Rise or fall of Vitamin E after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- Vitamin B1 (Active Comparator): Rise or fall of Vitamin B1 after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- Vitamin B2 (Active Comparator): Rise or fall of Vitamin B2 after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- Vitamin B6 (Active Comparator): Rise or fall of Vitamin B6 after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- Vitamin B12 (Active Comparator): Rise or fall of Vitamin B12 after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- Vitamin C (Active Comparator): Rise or fall of Vitamin C after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- Vitamin D (Active Comparator): Rise or fall of Vitamin D after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- Calcium (Active Comparator): Rise or fall of Calcium after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- Iron (Active Comparator): Rise or fall of Iron after three months
  Interventions: Dietary Supplement: EZPAK; Dietary Supplement: Placebo
- IGF1 (No Intervention): Rise or fall of IGF1 after three months
- FT-3 (No Intervention): Rise or fall of FT-3 after three months

INTERVENTIONS:
Dietary Supplement: EZPAK — One packet with breakfast for three months
  Arms: Calcium; Iron; Vitamin A; Vitamin B1; Vitamin B12; Vitamin B2; Vitamin B6; Vitamin C; Vitamin D; Vitamin E
Dietary Supplement: Placebo — One packet with breakfast for three months
  Arms: Calcium; Iron; Vitamin A; Vitamin B1; Vitamin B12; Vitamin B2; Vitamin B6; Vitamin C; Vitamin D; Vitamin E

SUMMARY:
The purpose of this study is to correlate the findings of an early study with current data.

ELIGIBILITY:
Inclusion Criteria: Healthy volunteers whose circulating serum vitamin A1, E, B1,B2,B6,B12,C,D, Calcium, Iron, IGF-1 and FT-3 are within normal limits.

A1; 48-85 ug/dl, E; 5.3-17.5 mg/L, B1; 66.5-200 nmo/L, B2; 137-370 ug/L, B6; 2-32.8 ug/L, B12; 211-946 pg/mL, C; 0.2-2.0 mg/dL, D; 30-100 ng/mL, Calcium; 8.7-10.2 mg/dL, Iron; 27-159 ug/dL, IGF-1; 67-205 ng/mL, FT-3; 2-4.4 pg/mL

Exclusion Criteria: Volunteers whose circulating serum vitamin A1, E, B1,B2,B6,B12,C,D, Calcium, Iron, IGF and FT-3 are outside normal limits.

A1; 48-85 ug/dl, E; 5.3-17.5 mg/L, B1; 66.5-200 nmo/L, B2; 137-370 ug/L, B6; 2-32.8 ug/L, B12; 211-946 pg/mL, C; 0.2-2.0 mg/dL, D; 30-100 ng/mL, Calcium; 8.7-10.2 mg/dL, Iron; 27-159 ug/dL, IGF-1; 67-205 ng/mL, FT-3; 2-4.4 pg/mL -

Ages: 26 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Raise in Circulating Serum Vitamin A1, E, B1,B2,B6,B12,C,D, Calcium, Iron, IGF and FT-3. | Three months
  Effectiveness of EZPAK in Raising Circulating Serum Levels

SECONDARY OUTCOMES:
Control group | Three months
  Levels of Circulating Serum VitaminA1, E, B1,B2,B6,B12,C,D, Calcium, Iron, IGF and FT-3.
Placebo group | Three months
  Levels of Circulating Serum VitaminA1, E, B1,B2,B6,B12,C,D, Calcium, Iron, IGF and FT-3.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Osguthorpe, ND, Principal Investigator — Optimal Health Research
Locations (1):
- Optimal Health Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nenseth HZ, Sahu A, Saatcioglu F, Osguthorpe S. A Nutraceutical Formula Is Effective in Raising the Circulating Vitamin and Mineral Levels in Healthy Subjects: A Randomized Trial. Front Nutr. 2021 Sep 1;8:703394. doi: 10.3389/fnut.2021.703394. eCollection 2021. PMID 34540877